CLINICAL TRIAL: NCT05579132
Title: An Open-label, Multi-center Phase Ib/II Study of MK-1045 (CN201) in Subjects With Precursor B-cell Acute Lymphoblastic Leukemia
Brief Title: A Clinical Study of MK-1045 (CN201) in People With Precursor B-cell Acute Lymphoblastic Leukemia (MK-1045-002)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MSD R&D (China) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1045-002; MK-1045-002 (Other: MSD); CN201-103 (Other: Curon Biopharmaceutical Co., LTD)
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MK-1045: Dose Escalation Phase- Adult Cohort (Experimental): Adults in the dose escalation phase will receive a target dose level of MK-1045 from 600 μg to 90000 μg, administered by intravenous (IV) infusion. MK-1045 will be administered once per week, in treatment cycles defined as 4 weeks of MK-1045 treatment.
  Interventions: Drug: MK-1045
- MK-1045 : Dose Escalation Phase- Pediatric Cohort (Experimental): Pediatric participants will receive a target dose level of MK-1045 from 320 μg to 60000 μg, with dosing further based upon weight. MK-1045 will be administered by IV infusion once per week, in treatment cycles defined as 4 weeks of MK-1045 treatment.
  Interventions: Drug: MK-1045

INTERVENTIONS:
Drug: MK-1045 — MK-1045 is administered by IV infusion once a week (QW), 4 weeks per treatment cycle, starting with 2 cycles of induction treatment. After a 2-week treatment-free interval, responders to induction treatment receive 3 cycles of consolidation therapy, and up to 7 cycles of maintenance treatment or until intolerable toxicity, disease progression, withdrawal of informed consent, loss to follow-up, receipt of other antitumor therapy, or death, whichever occurs first. Each 4 week treatment cycle is followed by a 2-week treatment-free interval
  Other Names: CN201

SUMMARY:
Researchers are looking for new ways to treat people with a type of blood cancer called precursor B-cell Acute Lymphoblastic Leukemia (B-ALL) that is relapsed- the cancer has come back after treatment, or refractory - the current treatment has stopped working to slow or stop cancer growth. This study will have two parts. In the first part (dose escalation phase) the goal is to learn about the safety of a study treatment, MK-1045, and to find the best dose level of MK-1045 that is tolerated and may work to treat B-ALL. In the second part (Phase II) researchers want to learn how well MK-1045 works to treat B-ALL

ELIGIBILITY:
The main inclusion criteria include but are not limited to:

* Adult participants must be age 18 or older
* Pediatric participants must be at least 2 years old and less than 18 years old.
* Diagnosis of precursor B-cell acute lymphoblastic leukemia (B-ALL) and have more than 5% blasts in the bone marrow by morphological assessment
* Participants with Ph-negative B-ALL with any of the following refractory/relapse criteria:

  * Failure to achieve complete remission after initial induction therapy;
  * Failure to achieve complete remission after salvage treatment;
  * Relapse with first remission duration ≤12 months
  * Second or later relapse
  * Relapse after allogeneic HSCT
* Participants with Ph-positive B-ALL who have received 2 (or more) tyrosine kinase inhibitors (TKIs) and meet the refractory/relapse criteria above or, those with the T315I mutation

The main exclusion criteria include but are not limited to:

* History of Burkitt's leukemia.
* Received anti-CD19 therapy within 3 months prior to entering the study
* Received allogeneic HSCT within 12 weeks prior to entering the study
* Received prior treatment with chimeric antigen receptor T cell (CAR-T) within 3 months prior to entering the study
* History or presence of clinically relevant central nervous system (CNS) pathology
* History of clinically symptomatic metastases to the central nervous system or meninges, or other evidence of uncontrolled metastases to the CNS or meninges
* History of immunodeficiency, including history of any positive test result for human immunodeficiency virus (HIV) antibody.
* History of serious cardiovascular and cerebrovascular disease
* Has active autoimmune diseases that may relapse

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase: Number of Participants who Experience at Least One Adverse Event (AE) | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Dose Escalation Phase: Number of Participants who Discontinue Study Treatment Due to an AE | Up to approximately 21 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Dose Escalation Phase: Number of Participants Who Experience a Dose-limiting Toxicity (DLT) | Up to 28 days
  A DLT is defined as any of the following toxicities and judged by the investigator to be related to the study drug:
  Hematologic toxic reactions: If thrombocytopenia, leukopenia, and anemia are caused by primary leukemia, they are not considered as DLTs.
  Non-Hematologic toxic reactions: Grade 4 non-hematologic toxicity that does not recover to ≤ Grade 2 within 14 days of best supportive therapy. Grade 3 rash, fatigue, fever, or infection will not be classified as DLT; other Grade 3 non-hematologic toxicities that do not recover to ≤ Grade 2 within 14 days of best supportive therapy is considered DLTs.
  Others that are considered as DLTs: Other toxicities considered clinically significant by the investigator that result in permanent drug withdrawal.
Dose Escalation Phase: Maximum Tolerated Dose (MTD) of MK-1045 | Up to approximately 21 months
  The MTD will be determined based on the incidence of DLT in each dose level. The dose level for which the DLT rate is closest to the target DLT rate (30%) will be selected as the MTD.
Phase II: Complete Remission (CR) Rate | Up to approximately 10 weeks
  Complete remission is defined as follows:
  < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L. The number of participants with CR will be presented.

SECONDARY OUTCOMES:
Dose Escalation Phase: Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of MK-1045 | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the AUC from time 0 to the last concentration that can be accurately measured of MK-1045
Dose Escalation Phase: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of MK-1045 | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the AUC0-inf of MK-1045.
Dose Escalation Phase: Area Under the Concentration-time Curve From Time 0 to 168 hours (AUC0-168) | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the AUC from time to 168 hours after the start of infusion of MK-1045
Dose Escalation Phase: AUC From Time 0 to 168 Hours at Steady State (AUC0-tau) | At designated time points up to 24 weeks
  Blood samples will be collected to determine the AUC0 -tau
Dose Escalation Phase: Maximum Serum Drug Concentration (Cmax) of MK-1045 | At designated time points up to approximately 32 weeks
  Blood samples will be collected to determine the maximum serum drug concentration, obtained directly from the measured value of the plasma concentration-time curve
Dose Escalation Phase: Time to Maximum Serum Drug Concentration of MK-1045 | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the Tmax of MK-1045
Dose Escalation Phase: Concentration at End of Dosing Interval (Ctrough) of MK-1045 | At designated time points up to approximately 12 months
  Blood samples will be collected to determine the Ctrough of MK-1045
Dose Escalation Phase: Apparent Terminal Half Life (t1/2) | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the t1/2 of MK-1045
Dose Escalation Phase: Apparent Clearance (CL) of MK-1045 | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the CL of MK-1045
Dose Escalation Phase: Apparent Volume of Distribution (Vz) of MK-1045 | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the Vz of MK-1045
Dose Escalation Phase: Apparent Volume of Distribution at Theoretical Steady State (Vss) of MK-1045 | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the Vss of MK-1045
Dose Escalation Phase: Mean Residence Time (MRT) of MK-1045 | At designated time points up to approximately 24 weeks
  Blood samples will be collected to determine the MRT of MK-1045
Dose Escalation Phase: Peripheral B Cell Depletion of MK-1045 | Baseline and at designated time points up to approximately 12 months
  B cell depletion will be determined at each timepoint by comparing absolute B cell numbers (as determined by flow cytometry) with those at baseline
Dose Escalation Phase: Peripheral Circulating T Cell Activation of of MK-1045 | Baseline and at designated time points up to approximately 12 months
  Peripheral circulating T cell activation will be determined at each timepoint by comparing absolute T cell numbers and T cell activation markers with those at baseline
Dose Escalation Phase: Percentage of Participants with Antidrug Antibodies (ADA) to MK-1045 | At designated time points up to approximately 12 months
  Blood samples collected at designated timepoints will be used to determine the percentage of participants who develop detectable ADAs to MK-1045
Dose Escalation Phase: Rate of Complete Remission (CR) and Complete Remission with Partial Hematologic Recovery (CRh) | Up to approximately 10 weeks
  Complete remission is defined as follows:
  < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L.
  CRh is defined as meeting all of the following criteria:
  Satisfaction of all criteria for CR except partial recovery of peripheral blood counts (platelets ≥ 50 ×10^9/L and ANC ≥ 0.5×10^9/L). The percentage of participants with CR or CRh will be presented.
Dose Escalation Phase: Rate of CR, CRh, and Complete Response with Incomplete Hematologic Recovery (CRi) | Up to approximately 10 weeks
  Complete remission is defined as follows:
  < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L.
  CRh is defined as meeting all of the following criteria:
  Satisfaction of all criteria for CR except partial recovery of peripheral blood counts (platelets ≥ 50 ×10^9/L and ANC ≥ 0.5×10^9/L).
  CRi is defined as follows:
  <5% blasts in the bone marrow, No circulating lymphoblasts or extramedullary disease, and platelets <100×10^9/L and neutrophils ≥1.0×109/L or platelets ≥100 ×109/L and neutrophils <1.0×10^9/L. The percentage of participants with CR, CRh or CRi will be presented.
Dose Escalation Phase: Rate of Minimum Residual Disease (MRD)-negative Complete Remission | Up to approximately 12 months
  MRD-negative is defined as less than 0.01% of leukemic cells were detected in bone marrow with a detection sensitivity no less than 10^-4.
Dose Escalation Phase: Rate of Red Blood Cell and Platelet Transfusion Independence (TI) | Up to approximately 24 months
  TI is defined as no transfusion for a period of at least 1 week (7 days). The percentage of participants having TI will be presented.
Phase II: Number of Participants Who Experience at Least 1 AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Phase II: Number of Participants who Discontinue Study Treatment Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Phase II: Maximum Serum Drug Concentration (Cmax) of MK-1045 | At designated time points up to 4 weeks
  Blood samples will be collected to determine the maximum serum drug concentration, obtained directly from the measured value of the plasma concentration-time curve
Phase II: Concentration at End of Dosing Interval (Ctrough) of MK-1045 | At designated time points up to 4 weeks
  Blood samples will be collected to determine the Ctrough of MK-1045
Phase II: Peripheral B Cell Depletion of MK-1045 | Baseline and at designated time points up to 4 weeks
  B cell depletion will be determined at each timepoint by comparing absolute B cell numbers (as determined by flow cytometry) with those at baseline
Phase II: Peripheral Circulating T Cell Activation of of MK-1045 | Baseline and at designated time points up to 4 weeks
  Peripheral circulating T cell activation will be determined at each timepoint by comparing absolute T cell numbers and T cell activation markers with those at baseline
Phase II: Concentration of Peripheral Cytokines | Baseline and at designated time points up to 4 weeks
  Blood samples will be collected to compare peripheral blood cytokine levels at various time points with those at baseline
Phase II: Percentage of participants with Antidrug Antibodies (ADA) to MK-1045 | At designated time points up to 4 weeks
  Blood samples collected at designated timepoints will be used to determine the percentage of participants who develop detectable ADAs to MK-1045
Phase II: Rate of CR and CRh | Up to approximately 10 weeks
  Complete remission is defined as follows:
  < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L.
  CRh is defined as meeting all of the following criteria:
  Satisfaction of all criteria for CR except partial recovery of peripheral blood counts (platelets ≥ 50 ×10^9/L and ANC ≥ 0.5×10^9/L). The percentage of participants with CR or CRh will be presented.
Phase II: Rate of CR/CRh/CRi | Up to approximately 10 weeks
  CR is defined as follows:
  < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L.
  CRh is defined as meeting all of the following criteria:
  Satisfaction of all criteria for CR except partial recovery of peripheral blood counts (platelets ≥ 50 ×10^9/L and ANC ≥ 0.5×10^9/L).
  CRi is defined as follows:
  <5% blasts in the bone marrow, No circulating lymphoblasts or extramedullary disease, and platelets <100×10^9/L and neutrophils ≥1.0×109/L or platelets ≥100 ×109/L and neutrophils <1.0×10^9/L. The percentage of participants with CR, CRh or CRi will be presented.
Phase II: Rate of Minimum Residual Disease (MRD)-negative Complete Remission | Up to approximately 24 months
  MRD-negative is defined as less than 0.01% of leukemic cells were detected in bone marrow with a detection sensitivity no less than 10^-4.
Phase II: Rate of Red Blood Cell and Platelet TI | Up to approximately 24 months
  Red Blood Cell and Platelet TI is defined as no transfusion for a period of at least 1 week (7 days). The percentage of participants having TI will be presented.
Phase II: Proportion of Participants Undergoing Hematopoietic Stem Cell Transplantation (HSCT) | Up to approximately 24 months
  The number of participants who undergo a HSCT during study participation will be presented.
Phase II: Duration of CR | Up to approximately 24 months
  For participants who demonstrate a CR (defined as < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L) , duration of CR is defined as the time from the first documentation of a disease response of CR to the date of the first documented relapse event, or death due to any cause, whichever occurs first
Phase II: Duration of CR/CRh | Up to approximately 24 months
  Duration of CR/CRh is defined as the time from the first documentation of a disease response of CR/CRh to the date of the first documented relapse event, or death due to any cause, whichever occurs first. Only participants who demonstrate a CR (defined as < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L), or CRh [satisfaction of all criteria for CR except partial recovery of peripheral blood counts (platelets ≥ 50 ×10^9/L and ANC ≥ 0.5×10^9/L)] will be analyzed.
Phase II: Duration of CR/CRh/CRi | Up to approximately 24 months
  Duration of CR/CRh/CRi is defined as the time from the first documentation of a disease response of CR/CRh/CRi to the date of the first documented relapse event, or death due to any cause, whichever occurs first. Only participants who demonstrate a CR (defined as < 5% blasts in the bone marrow, no circulating lymphoblasts or extramedullary disease, and full recovery of peripheral blood counts: Platelets ≥100×10^9/L, and absolute neutrophil count (ANC) ≥1.0×10^9/L), or CRh [satisfaction of all criteria for CR except partial recovery of peripheral blood counts (platelets ≥ 50 ×10^9/L and ANC ≥ 0.5×10^9/L)], or CRi (<5% blasts in the bone marrow, No circulating lymphoblasts or extramedullary disease, and platelets <100×10^9/L and neutrophils ≥1.0×109/L or platelets ≥100 ×109/L and neutrophils <1.0×10^9/L) will be analyzed.
Phase II: Relapse-Free Survival (RFS) | Up to approximately 24 months
  RFS is defined as the time from the first dose of MK-1045 to the first documented relapse, or death due to any cause (whichever occurs first). In participants who achieve CR, CRh or CRi, relapse is defined as either hematological or extramedullary relapse . Hematological relapse is defined as recurrence of blasts in the blood, or >5% blasts in bone marrow. Extramedullary relapse is defined as recurrence of extramedullary disease after a CR.
Phase II: Overall Survival (OS) | Up to approximately 24 months
  OS is the time from date of first study treatment to the date of death due to any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (11):
- China (11):
  - The Second Affiliated Hospital of Third Military Medical University ( Site 0008), Chongqing, Chongqing Municipality
  - Southern Medical University Nanfang Hospital ( Site 0004), Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University ( Site 0003), Shijiazhuang, Hebei
  - The First Hospital of Harbin ( Site 0005), Harbin, Heilongjiang
  - Henan Cancer Hospital-hematology department ( Site 0002), Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology ( Site 0010), Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of HUST ( Site 0006), Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University ( Site 0007), Xuzhou, Jiangsu
  - West China Second University Hospital, Sichuan University ( Site 0011), Chengdu, Sichuan
  - Hematology Hospital of Chinese Academy of Medical Sciences ( Site 0001), Tianjin, Tianjin Municipality
  - The Children's Hospital of Zhejiang University School of Medicine ( Site 0009), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com